CLINICAL TRIAL: NCT04536272
Title: Reduced Anticoagulation Targets in ECLS (RATE)
Acronym: RATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Erasmus Medical Center (Other); Leiden University Medical Center (Other); St. Antonius Hospital (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Isala (Other); OLVG (Network); Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Walter M. van den Bergh, Principal investigator, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201900659; 848018014 (Other Grant/Funding Number: ZonMW); 7969 (Registry Identifier: Netherlands Trial Register); 2019-004125-24 (EudraCT Number)
Record Dates: First submitted 2020-08-24; First posted 2020-09-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure; Respiratory Failure; Extracorporeal Membrane Oxygenation; Bleeding; Thrombosis
Keywords: Extracorporeal membrane oxygenation; Extracorporeal life support; ECMO; ECLS; Anticoagulation; Complications
MeSH Terms: conditions — Heart Failure; Respiratory Insufficiency; Hemorrhage; Thrombosis | interventions — Heparin; Heparin, Low-Molecular-Weight; Enoxaparin; Nadroparin

STUDY DESIGN:
Intervention Model Description: Randomization between anticoagulation targets during ECLS of: 1). 2-2.5 times baseline aPTT (usual care, about 60-75 sec.), 2). 1.5-2.0 times baseline aPTT (45-60 sec.) or 3). LMWH guided by weight and renal function.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Target of 2-2.5 times baseline aPTT (usual care, about 60-75) (Active Comparator): Administration of heparin during ECLS with an aPTT target of 2-2.5 times baseline.
  Interventions: Drug: Heparin
- Target of 1.5-2.0 times baseline aPTT (45-60 sec.) (Active Comparator): Administration of heparin during ECLS with an aPTT target of 1.5-2.0 times baseline.
  Interventions: Drug: Heparin
- LMWH guided by weight and renal function. (Active Comparator): Administration of LMWH guided by weight and renal function during ECLS.
  Interventions: Drug: LMWH

INTERVENTIONS:
Drug: Heparin — Administration of heparin with a target of 2-2.5 or 1.5-2.0 times baseline aPTT during ECLS.
  Other Names: Unfractionated heparin
  Arms: Target of 1.5-2.0 times baseline aPTT (45-60 sec.); Target of 2-2.5 times baseline aPTT (usual care, about 60-75)
Drug: LMWH — Administration of LMWH guided by weight and renal function during ECLS.
  Other Names: Dalteparine; Enoxaparine; Nadroparine; Tinzaparine
  Arms: LMWH guided by weight and renal function.

SUMMARY:
The objective of the RATE-trial is to study if reduced anticoagulation targets during ECLS diminish bleeding complications without an increase in thromboembolic complications or a negative impact on outcome.

DETAILED DESCRIPTION:
Rationale: ECMO treatment has a mortality of 38%, for a large part treatment related due to complications. The most feared complication is ischemic stroke for which heparin is administered with an aPTT target 2.0-2.5 times baseline (approximately 60-75 sec).

However, there is no relation between aPTT and the occurrence of stroke (1.2%), but there is a relation with the much more frequent occurrence of bleeding complications (55%) and blood transfusion. Both are strongly related to outcome.

Objective: Our objective is to study if reduced anticoagulation targets diminish bleeding complications without an increase in thromboembolic complications or a negative impact on outcome.

Study design: Three-arm non-inferiority RCT.

Study population: All adult Dutch patients treated with ECMO during the 30 months of the study.

Intervention: Randomization between heparin administration with a target of 2-2.5 times baseline aPTT (usual care, about 60-75 sec.), 1.5-2.0 times baseline aPTT (45-60 sec.) or low molecular weight heparin (LMWH) guided by weight and renal function.

Main study parameters/endpoints: The primary outcome parameter is a combined endpoint consisting of: 1) major bleeding including hemorrhagic stroke according to the ELSO definitions; 2) severe thromboembolic complication defined as ischemic stroke, limb ischemia (not related with distal perfusion catheter), or acute pump failure with emergency exchange; 3) mortality at 6 months.

Secondary outcome parameters are: 1) blood transfusions; 2) health related quality of life (HR-QoL) at 6 months; 3) exchange of the membrane oxygenator; 4) vessel thrombosis after ECMO removal detected by echography; 5) pulmonary embolism; 6) costs; 7) the individual components of the composite outcome; and 8) all thromboembolic complications combined.

Expected outcomes: We expect that with a target of 1.5-2.0x baseline aPTT or with LMWH the primary composite endpoint will be reached in 60% of patients compared to 70% in usual care. To show non-inferiority with a significance level (alpha) of 5%, power of 80% and a non-inferiority limit (delta) of 7.5% the corresponding sample size is 91 patients per group. In other words, if there is a true difference in favor of the experimental treatment of 10%, then 91 patients per group are required to be 80% sure that the upper limit of a one-sided 95% confidence interval (or equivalently a 90% two-sided confidence interval) will exclude a difference in favor of the standard group of more than 7.5%. To compensate for a lower effect and drop-outs 330 patients will be enrolled. Apart from anticoagulation targets, treatment will be as usual so study participation will not lead to a burden for the patient, e.g. no extra blood sampling, tests or visits. After 6 months the patients will be contacted for a short questionnaire to measure health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* ECMO treatment during the study period in one of the participating centers
* Age above 18 years
* Written informed consent

Exclusion Criteria:

* Patients in whom the ECMO is only used to bridge a procedure
* Vital indication for robust anticoagulation (e.g. mechanic valve, pulmonary embolism)
* History of heparin induced thrombocytopenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-03-07 (Actual)

PRIMARY OUTCOMES:
Hemorrhagic complications | Through ECLS completion, an average of 14 days
  Severe hemorrhagic complications will be registered according to the Extracorporeal Life Support Organization (ELSO) definitions for major bleeding and is defined as clinically overt bleeding with a decrease in hemoglobin of at least 1,24 mmol/L (2 g/dl)/24 hours, or a transfusion requirement of ≥ 3 EH RBC over that same time period. Bleeding that is retroperitoneal, pulmonary or involves the central nervous system, or bleeding that requires surgical intervention is also considered major bleeding.
Severe thromboembolic complications | Through ECLS completion, an average of 14 days
  Severe thromboembolic complication defined as ischemic stroke, limb ischemia, or acute pump failure
Mortality | 6 months after ECLS
  Mortality at 6 months

SECONDARY OUTCOMES:
Number of blood transfusions | Through ECLS completion, an average of 14 days
  Number of blood transfusions during ECLS
Quality of life at 6 months | 6 months after ECLS
  Quality of life (HR-QoL) measured 6 months after decannulation from ECMO
Exchange of the membrane oxygenator | Through ECLS completion, an average of 14 days
  Number of echanges of the membrane oxygenator during ECLS
Vessel thrombosis after ECLS removal | After ECLS completion, an average of 14 days
  Vessel thrombosis after ECLS removal detected by echography
Cost- effectiveness | 6 months after ECLS
  Cost- effectiveness will be based on reduced costs of blood transfusions and interventions for bleeding (e.g. surgery, interventional radiology) as well as improved outcome. All medical cost items expected to be affected by the ECMO therapy will be measured and valued according to the Dutch standard guidelines for economic evaluations, e.g. blood transfusion, number of ECMO replacements, surgery, and hospital length of stay.
Pulmonary embolism | Through ECLS completion, an average of 14 days
  The occurrence of Pulmonary embolism during ECLS
All thromboembolic complications combined | Through ECLS completion, an average of 14 days
  The occurrence of all thromboembolic complications combined during ECLS

CONTACTS AND LOCATIONS:
Overall Officials: W.M. van den Bergh, PhD, MD, Principal Investigator — University Medical Center Groningen
Locations (8):
- Netherlands (8):
  - Radboud UMC, Nijmegen, Gelderland
  - Maastricht Universitair Medisch Centrum+, Maastricht, Limburg
  - OLVG, location East, Amsterdam, North Holland
  - Amsterdam UMC, location AMC, Amsterdam, North Holland
  - Isala Clinics, Zwolle, Overijssel
  - University Medical Center Groningen, Groningen, Provincie Groningen
  - Leids Universitair Medisch Centrum, Leiden, South Holland
  - Erasmus MC, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: * Researchers who provide a methodologically sound proposal which is approved by an independent review panel.
  * To achieve aims in the approved proposal.
  * Proposals should be directed to w.m.van.den.bergh@umcg.nl, requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] van Minnen O, Linde M, Oude Lansink-Hartgring A, van den Boogaard B, Bunge JJH, Delnoij TSR, Elzo Kraemer CV, Kuijpers M, Maas JJ, de Metz J, van de Poll M, Dos Reis Miranda D, Vlaar APJ, van Ravenzwaaij D, van den Bergh WM. Reduced anticoagulation targets in extracorporeal life support (RATE): protocol for a pre-planned secondary Bayesian analysis of the rate trial. Trials. 2025 Mar 15;26(1):90. doi: 10.1186/s13063-025-08737-6. PMID 40087802
- [Derived] van Minnen O, Oude Lansink-Hartgring A, van den Boogaard B, van den Brule J, Bulpa P, Bunge JJH, Delnoij TSR, Elzo Kraemer CV, Kuijpers M, Lambermont B, Maas JJ, de Metz J, Michaux I, van de Pol I, van de Poll M, Raasveld SJ, Raes M, Dos Reis Miranda D, Scholten E, Simonet O, Taccone FS, Vallot F, Vlaar APJ, van den Bergh WM. Reduced anticoagulation targets in extracorporeal life support (RATE): study protocol for a randomized controlled trial. Trials. 2022 May 16;23(1):405. doi: 10.1186/s13063-022-06367-w. PMID 35578271